CLINICAL TRIAL: NCT06229587
Title: Speech and Middle Ear Outcomes Following Primary Cleft Palate Repair by Furlow Z-plasty Technique With a Buccinator Myomucosal Flap
Brief Title: Furlow With Buccinator and Velopharyngeal Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohsen, principle investigator, Fayoum University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13
Record Dates: First submitted 2024-01-01; First posted 2024-01-29 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Cleft Palate
MeSH Terms: conditions — Cleft Palate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- furlow with buccinator arm (Experimental)
  Interventions: Procedure: furlow with buccinator flap

INTERVENTIONS:
Procedure: furlow with buccinator flap — Assessment of speech and the middle ear function of patients between the age of 3 and 7 years surgically treated by ARC (Furlow z-palatoplasty with a buccinator myomucosal flap) was done

SUMMARY:
Assessment of speech and the middle ear function of patients between the age of 3 and 7 years surgically treated by ARC (Furlow z-palatoplasty with a buccinator myomucosal flap) was done. Middle ear function was assessed by clinical otoscopic examination and by tympanometry to detect the presence or absence of middle ear effusion and the need for tympanostomy tubes. Speech outcomes were assessed using perceptual speech assessment for the degree of hypernasality, compensatory misarticulation and speech intelligibility. Nasopharyngoscopic examination of the patients was done for visualization of the velopharyngeal port, allowing assessment of the pattern and grade of velopharyngeal closure during speech and the presence or absence of a velopharyngeal gap

ELIGIBILITY:
Inclusion Criteria:

* - Age 3 to 7 years
* 1ry cleft repair by furrolow with buccal myomucosal flap
* Non syndromic previously treated children
* Cleft repaired by the same surgeon

Exclusion Criteria:

* - Syndromic patient
* Cleft palate repair by any technique except furlow with buccal myomucosal flap

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
speech assessement | 3years
  Nasopharyngoscopic examination of the cleft patients after repair with Furlow with buccinator flap allowing assessment of the grade of velopharyngeal closure during speech

CONTACTS AND LOCATIONS:
Locations (1):
- Hearing Institution, Giza, Egypt